CLINICAL TRIAL: NCT06228612
Title: How Far Are Vacuum Therapy and Stabilization Splints Efficacious for the Management of Temporo-mandibular Joint Osteoarthritis? A Randomized Clinical Trial.
Brief Title: Vacuum Therapy and Stabilization Splints Efficacious for the Management of Temporo-mandibular Joint Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A12060922
Record Dates: First submitted 2023-12-13; First posted 2024-01-29 (Actual); Last update posted 2024-01-29 (Actual); Status verified 2020-12

CONDITIONS: Osteoarthritis
Keywords: TMJ, osteoarthritis, vacuum, stabilization splint.
MeSH Terms: conditions — Osteoarthritis | interventions — Negative-Pressure Wound Therapy

STUDY DESIGN:
Intervention Model Description: Patient's randomization was performed by two assistants who did not participate in the trial. One assistant had prepared sequentially numbered sealed envelopes with random assignment. The assignment of the treatment was then completed by another assistant from outside the trial. Patients whose treatment plans included vacuum therapy (VT) were designated group (I) and included 14 patients, and those with stabilization splint therapy (SST) were designated (group (II) and included 14 patients. Patients whose treatment plans included both vacuum therapy and splint therapy (VT + SST) were designated as group (III) and included 14 patients.
Who Masked: Participant, Outcomes Assessor
Masking Description: Patient's randomization was performed by two assistants who did not participate in the trial. One assistant had prepared sequentially numbered sealed envelopes with random assignment. The assignment of the treatment was then completed by another assistant from outside the trial.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- group I:vacuum therapy (Active Comparator): group I:vacuum therapy VT:patients who were diagnosed with TMJ osteoarthritis. The patients received Isolated vacuum therapy VT
  Interventions: Device: vacuum therapy
- group II: maxillary stabilization splint (MSS) (Active Comparator): group II, patients who were diagnosed with TMJ osteoarthritis. The patients received stabilization splint therapy (STT)
  Interventions: Device: maxillary stabilization splint (MSS)
- group III: vacuum therapy VT and maxillary stabilization splint (MSS) (Active Comparator): group III: patients who were diagnosed with TMJ osteoarthritis. The patients received combined VT and SST.
  Interventions: Device: vacuum therapy VT and maxillary stabilization splint (MSS)

INTERVENTIONS:
Device: vacuum therapy — vacuum therapy :all patients were informed about initial suction sensation and possible appearance of bruising at the application site. Basic vacuum therapy equipment (cangexia, China) was utilized including a manual suction pump, plastic cups of 40 mm diameter with rolled edge, and anti-septic tools.
  Arms: group I:vacuum therapy
Device: maxillary stabilization splint (MSS) — maxillary stabilization splint (MSS): was constructed for each patient from hard, heat-cured clear acrylic resin and fitted to the maxillary teeth. On the mounted master casts, the vertical dimension was adjusted to provide 3 mm of vertical space between the closest opposing cusps of the maxillary and mandibular teeth.
  Arms: group II: maxillary stabilization splint (MSS)
Device: vacuum therapy VT and maxillary stabilization splint (MSS) — vacuum therapy VT and maxillary stabilization splint (MSS): both Basic vacuum therapy and maxillary stabilization splint :Procedures were the same as in group I and II.
  Arms: group III: vacuum therapy VT and maxillary stabilization splint (MSS)

SUMMARY:
The aim of this study was to determine and compare the clinical efficacy of VT and STT alone or in combination for the patients with temporo-mandibular joint (TMJ) osteoarthritis.

DETAILED DESCRIPTION:
Study design and patients´ selection:

This prospective parallel randomized clinical trial included patients diagnosed with TMJ osteoarthritis. All Patients were collected from the TMD clinic of Prosthodontics Department, Faculty of Dentistry, Mansoura University. The study was approved by the local ethics committee with ethical approval number A12060922. All patients were aware of the treatment procedures and signed informed consents for their participation. Patients were recruited and data collection was performed between . CONSORT guidelines were followed when approperiate19 Inclusion and exclusion criteria were defined prior to the beginning of the study. Inclusion criteria were: (I) clinical diagnosis of TMJ osteoatrhritis according to diagnostic criteria involved in the DC/TMD axis I group 3.A.2 item20 including self-report of TMJ pain, tenderness to palpation, and crepitus (II) magnetic resonance imaging (MRI)signs of joint effusion, erosions and ⁄ or sclerosis of the cortical outline, flattening of the joint surfaces and ⁄ or osteophyte formation ; and (III) age cognitively capable of understanding the standardized questionnaire.

Exclusion criteria were: (I) Patients with systemic disease affecting the joints (II) previous TMJ treatment, (III) previous trauma to TMJ or to the jaws, and (IV) edentulous patients, (V) use of anti-inflammatory drugs at least one month before assessment and during the treatment period.

Sample size calculation:

Sample size calculation was performed by using G*Power software (version 3.1.9.7) based on previous study by El-Shaheed et al.21 A medium effect size (f = 0.25) for interaction effect of treatment group and time on quantitative outcomes (amount of mouth opening in mm, temporo-mandibular joint palpation and VAS score for pain) and a large effect size (f = 0.4) for main group effect on these outcome measures were hypothesised. Based on these assumptions, a total sample size of 42 (14 in each treatment group) achieved 83% power to detect a large effect size (f = 0.4) with 0.05 α-error probability using F test anova: Repeated measures, between factors for three groups and five measurements with a .5 correlation between measurements.

Patients' randomization:

Patients who are eligible in this study after screening phase and who agree to sign the consent form were randomly assigned to grouping. Patient's randomization was performed by two assistants who did not participate in the trial. One assistant had prepared sequentially numbered sealed envelopes with random assignment. The assignment of the treatment was then completed by another assistant from outside the trial. Patients whose treatment plans included vacuum therapy (VT) were designated group (I) and included 14 patients, and those with stabilization splint therapy (SST) were designated (group (II) and included 14 patients. Patients whose treatment plans included both vacuum therapy and splint therapy (VT + SST) were designated as group (III) and included 14 patients.

Intervention:

The treatments were applied by an experienced dentist, with the necessary training in TMD specialty.

For group (I) (VT group), vacuum therapy was applied over the TMJ. Before intervention, all patients were informed about initial suction sensation and possible appearance of bruising at the application site. Basic vacuum therapy equipment (cangexia, China) was utilized including a manual suction pump, plastic cups of 40 mm diameter with rolled edge, and anti-septic tools. The cup can be fixed by means of fixation gel () before application of the cup as hair might interfere with the cup peripheral seal. Dry vacuum therapy was accomplished by application of constant negative pressure of 300 mbar (which is equal to two suctions) using the manual suction pump through the suction cup over the TMJ region for 5 minutes22 (Fig.1). Whether any extra oral muscle showed pain, vacuum therapy application was performed using the same protocol. After completing the procedures, an anti-septic solution was placed over the vacuum application site (sites). All patients in this group were treated one session per week for four successive weeks (Fig.2).

For group (II) (ST group), A maxillary stabilization splint (MSS) was constructed for each patient from hard, heat-cured clear acrylic resin and fitted to the maxillary teeth. On the mounted master casts, the vertical dimension was adjusted to provide 3 mm of vertical space between the closest opposing cusps of the maxillary and mandibular teeth. The occlusal contact of the splint was adjusted to provide even simultaneous contact with the opposing mandibular cusps in the treatment position. the mandibular canines provide laterotrusive guidance in lateral exertions (canine guidance), and mandibular anterior teeth provide anterior contact and posterior disocclusion (anterior guidance). After processing, the splint was fitted on the maxillary arch and adjusted if needed (Fig.3). Patients were advised to wear it 12 hours per day for six months. Patients were recalled regularly for occlusal readjustment of the splint.

For group (III) (VT+SST), both VT and SST were started at the same day. Procedures were the same as in group I and II.

Collagen hydrolysate

Patients' evaluation:

Patients' evaluation was performed by an experienced independent researcher who did not participate in other procedures in this study and was blinded to all intervention groups.

I- Clinical evaluation:

Patients were evaluated regarding their TMJ signs and symptoms at base line (T0), one week (Tw), one month (T1), three months (T3), and six months (T6):

1. Maximum comfortable mouth opening (MCO) was measured using millimeter ruler between the incisal edges plus the overbite while the patient opens at maximum comfortable opening.
2. The degree of pain was evaluated using 0 to10 mm Visual Analogue Scale (VAS) for pain (where 0 equals no pain and 10 is the most severe pain).
3. TMJ tenderness on palpation was assessed by Verbal Rating Scale (VRS) using firm and constant pressure of half kg lasted two seconds over the condyle in front of the tragus. The degree of joint tenderness was extended from 0 to 3 (0: no; 1: slight; 2: moderate; 3: severe).
4. Joint sound was detected using stethoscope
5. Change perception was assessed at Tw, T1, T3, and T6 with the Patient Global Impression of Change Scale (PGICS) which evaluates the change perceived by the patients after treatment. This scale has seven affirmations depicting a patient's rating of overall improvement (1 "very much improved", 2 "much improved", 3 "minimally improved", 4 "no change", 5 "minimally worse", 6 "much worse", or 7 "very much worse").
6. Any side effects from either treatments also had been reported.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria were: (I) clinical diagnosis of TMJ osteoatrhritis according to diagnostic criteria involved in the DC/TMD axis I group 3.A.2 item20 including self-report of TMJ pain, tenderness to palpation, and crepitus (II) magnetic resonance imaging (MRI)signs of joint effusion, erosions and ⁄ or sclerosis of the cortical outline, flattening of the joint surfaces and ⁄ or osteophyte formation ; and (III) age cognitively capable of understanding the standardized questionnaire.

Exclusion Criteria:

* Exclusion criteria were: (I) Patients with systemic disease affecting the joints (II) previous TMJ treatment, (III) previous trauma to TMJ or to the jaws, and (IV) edentulous patients, (V) use of anti-inflammatory drugs at least one month before assessment and during the treatment period.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2021-01-20 (Actual); Primary Completion 2022-12-03 (Actual); Study Completion 2023-11-17 (Actual)

PRIMARY OUTCOMES:
Maximum comfortable mouth opening (MCO), | 6 months
  Maximum comfortable mouth opening (MCO) was measured using millimeter ruler between the incisal edges plus the overbite while the patient opens at maximum comfortable opening.

SECONDARY OUTCOMES:
visual analogue scale (VAS), | 6 months
  The degree of pain was evaluated using 0 to10 mm Visual Analogue Scale (VAS) for pain (where 0 equals no pain and 10 is the most severe pain).

OTHER OUTCOMES:
Verbal Rating Scale (VRS) | 6 months
  TMJ tenderness on palpation was assessed by Verbal Rating Scale (VRS) using firm and constant pressure of half kg lasted two seconds over the condyle in front of the tragus. The degree of joint tenderness was extended from 0 to 3 (0: no; 1: slight; 2: moderate; 3: severe).
Patient Global Impression of Change Scale (PGICS), | 6 months
  Change perception was assessed at Tw, T1, T3, and T6 with the Patient Global Impression of Change Scale (PGICS) which evaluates the change perceived by the patients after treatment. This scale has seven affirmations depicting a patient's rating of overall improvement (1 "very much improved", 2 "much improved", 3 "minimally improved", 4 "no change", 5 "minimally worse", 6 "much worse", or 7 "very much worse").

CONTACTS AND LOCATIONS:
Overall Officials: Fatma Ahmad EL-Waseef, Associate professor, Principal Investigator — Faculty of Dentistry.Mansoura University,Prosthodontics Departement
Locations (1):
- Fatma A. EL Waseef, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: No